CLINICAL TRIAL: NCT07051369
Title: Frequency of Portal Hypertension Among Patient With Cirrhotic Liver With Ultrasound
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/920
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Portal Hypertension diagnostics — his study aims to determine the frequency of portal hypertension among patients with cirrhotic liver using ultrasound.A cross-sectional study will be conducted at Sheikh Zaid Medical College and Hospital, Rahim Yar Khan,

SUMMARY:
Portal hypertension is a common and serious complication of liver cirrhosis, often leading to life-threatening conditions such as variceal bleeding, ascites, and hepatic encephalopathy.

DETAILED DESCRIPTION:
Early detection and management are crucial for improving patient outcomes. While invasive methods such as hepatic venous pressure gradient (HVPG) measurement are the gold standard for diagnosis, they are costly and not widely available. Ultrasound, particularly Doppler imaging, offers a non-invasive, cost- effective alternative for assessing portal hypertension.This study aims to determine the frequency of portal hypertension among patients with cirrhotic liver using ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of chronic liver disease (CLD) will be included.
* Both male and female patients will be included.

Exclusion Criteria:

* Non-cirrhotic liver patients
* Non-cooperative patients.Patients who do not provide written informed consent

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: his study aims to determine the frequency of portal hypertension among patients with cirrhotic liver using ultrasound.A cross-sectional study will be conducted at Sheikh Zaid Medical College and Hospital, Rahim Yar Khan,
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Parameter Response | 12 Months
  this questioner will take the data from the ultrasound values having liver chirosis

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh Zayed college/hospital, Rahim Yar Khan, Punjab Province, Pakistan